CLINICAL TRIAL: NCT01795027
Title: A Prospective,Multicentral,Open-label,Randomized,Controlled,Phase III Clinical Trial to Compare S-1 Plus Oxaliplatin to S-1 as Adjuvant Chemotherapy After D2 Resection in Patients With Gastric Cancer
Brief Title: Compare S-1 Plus Oxaliplatin to S-1 as Adjuvant Chemotherapy After D2 Resection in Patients With Gastric Cancer
Acronym: CAPITAL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Zhiwei, Director of Gastric and Pancreatic Surgery,cancer center of Sun Yat-sen U, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCCGPS; ZHOUZHIWEI (Registry Identifier: ZZHIWEI)
Record Dates: First submitted 2013-02-14; First posted 2013-02-20 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; chemotherapy; D2 resection; S-1
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-1 plus Oxaliplatin (Experimental): 6 courses chemotherapy with S-1 plus oxaliplatin followed by 10 courses S-1 single after d D2 resection
  Interventions: Drug: S-1 plus oxaliplatin
- S-1 single (Active Comparator): S-1 40~60mg twice daily for 14 days in 3 weeks for totally 16 courses after D2 resection
  Interventions: Drug: S-1 single

INTERVENTIONS:
Drug: S-1 plus oxaliplatin — 6 courses chemotherapy with S-1 plus oxaliplatin followed by 10 courses S-1 single after d D2 resection
  Other Names: SOX
  Arms: S-1 plus Oxaliplatin
Drug: S-1 single — 16 courses S-1 single after d D2 resection
  Other Names: S-1
  Arms: S-1 single

SUMMARY:
Background: It is shown that TS-1 as adjuvant chemotherapy after D2 resection in patients with gastric cancer can improve DFS and OS in one Japanese Trial. And TS-1 has become one of the standard therapies to these patients. But it is still unknown whether it would improve more to OS and DFS than single TS-1 after combined with oxaliplatin . This trial is designed to investigate the efficacy and safety of TS-1 plus oxaliplatin versus TS-1 single as adjuvant chemotherapy after D2 resection in patients with gastric cancer.

Patients and methods: In this study , patients with histologically confirmed gastric cancer who received D2 resection and staged II or III, aged from 18 to 70 years and with Eastern Cooperative Oncology Group performance status ≤2 and adequate organ function, are randomized 1:1 to oxaliplatin 100mg/m2 on day 1 and TS-1 40~60mg twice everyday for 14 days in a 21-days cycle for total 6 cycles followed by TS-1 single with the same dose and frequency to the end of the 1st year postoperatively(SOX) , or TS-1 single 40~60mg twice everyday for 14 days in a 21-days cycle to the end of the 1st year postoperatively (TS-1). The primary end point is overall survival (OS), and secondary end point is disease free survival(DFS) and safety. Final study analysis will be conducted in the end of the 5th year after the last patient's enrollment.

ELIGIBILITY:
Inclusion Criteria:

* informed consensus of patients
* be able to receive oral administration
* from 18 to 70 years old
* be proven to be primary adenocarcinoma of gastric cancer and staged II or III by pathological evidences
* without other chemotherapy and/or radiation against to the disease
* normal function of other organs including heart,liver ,kidney and so on
* Eastern Cooperative Oncology Group performance status:0~2

Exclusion Criteria:

* history of other malignancy
* allergic reaction to S-1 or oxaliplatin
* be enrolling in other clinical trials
* abnormal GI tract function
* dysfunction of other organs
* female in pregnancy or lactation,or refuse to receive Contraception measures during chemotherapy
* other situation to be judged not adaptive to the study by investigators

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-11 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 year

SECONDARY OUTCOMES:
disease-free survival | 3 year
Number of Participants with Adverse Events | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhiwei Zhou, PHD, Study Chair — SunYat-sen University
Locations (13):
- China (13):
  - the central hospital of Chaozhou, Chaozhou, Guangdong
  - the 1st people's hospital of Foshan, Foshan, Guangdong
  - cancer center of Guangzhou medical college, Guangzhou, Guangdong
  - cancer center of Sun yat-sen University, Guangzhou, Guangdong
  - Guangdong Traditional Medical Hospital, Guangzhou, Guangdong
  - the 1st affliated hospital of Guangdong pharmacuetic college, Guangzhou, Guangdong
  - the 1St Affliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - the 6th affliated hospital of Sun-yat-sen University, Guangzhou, Guangdong
  - the 1st hospital of Shantou University, Shantou, Guangdong
  - the cental hospital of Shantou, Shantou, Guangdong
  - YUE-BEI people's hospital, Shaoguan, Guangdong
  - the 2nd people's hospital of Shenzhen, Shenzhen, Guangdong
  - the 5th hospital of Sun-yat-sen University, Zhuhai, Guangdong